CLINICAL TRIAL: NCT01969929
Title: Comparison of Postoperative Aqueous Flare After 20G Versus 23G Pars Plana Vitrectomy
Acronym: 20Gvs23G
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Sascha Fauser, MD, PhD, University of Cologne
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: UKK-13-247; 13-247 (Other: Ethics Committee University of Cologne)
Record Dates: First submitted 2013-10-18; First posted 2013-10-25 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Macular Hole; Macular Pucker
MeSH Terms: conditions — Retinal Perforations; Epiretinal Membrane | interventions — Vitrectomy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 20G (Active Comparator): 20G vitrectomy with scleral and conjunctival sutures for closure
  Interventions: Procedure: 20G Vitrectomy
- 23G (Active Comparator): 23G transconjunctival sutureless vitrectomy
  Interventions: Procedure: 23G vitrectomy

INTERVENTIONS:
Procedure: 20G Vitrectomy
  Arms: 20G
Procedure: 23G vitrectomy
  Arms: 23G

SUMMARY:
To compare postoperative inflammation and breakdown of blood-retinal barrier as measured by a laser flare-cell meter in 20G versus 23G vitrectomy.

ELIGIBILITY:
Inclusion Criteria:

age > 18 years macular hole macular pucker willing to perform follow up written signed consent

Exclusion Criteria:

other relevant eye disease: retinal detachment, provect cataract, diabetic retinopathy, AMD, relevant glaucoma, pre-surgery except for cataract surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-10; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Alteration of aqueous flare between preoperative and 3-week-postoperative time point | 3 weeks

SECONDARY OUTCOMES:
Visual acuity change | 3 weeks
Closure of Macular hole | 3 weeks

OTHER OUTCOMES:
Patient satisfaction | 3 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Center of Ophthalmology, University of Cologne, Cologne, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Scholz P, Muther PS, Schiller P, Felsch M, Fauser S. A Randomized Controlled Clinical Trial Comparing 20 Gauge and 23 Gauge Vitrectomy for Patients with Macular Hole or Macular Pucker. Adv Ther. 2018 Dec;35(12):2152-2166. doi: 10.1007/s12325-018-0826-6. Epub 2018 Nov 17. PMID 30448886